CLINICAL TRIAL: NCT04948411
Title: Durvalumab as Maintenance in Patients Who Received Chemoradiotherapy for Unresectable Stage III NSCLC: Real World Data From an Expanded Access Program in Brazil.
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 0120
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Durvalumab as maintenance in patients who received chemoradiotherapy for unresectable stage III NSCLC: Real World Data from an Expanded Access Program in Brazil

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable stage III NSCLC who completed a platinum-based chemotherapy concurrently or sequentially with radiation therapy without evidence of disease progression
2. Patients who have participated in the Durvalumab EAP in Brazil and have received at least one dose of Durvalumab in the EAP..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who have participated in the Durvalumab EAP in Brazil and have received at least 1 dose of Durvalumab.
  To enter the EAP, patients with unresectable stage III NSCLC must have completed a platinum-based chemotherapy concurrently or sequentially with radiation therapy without evidence of disease progression. It was preferred that treatment had started within approximately three months from end of radiation for patients to recover from treatment-related toxicities and/or for treating physicians to have adequate time to perform the baseline disease assessment. There was no fixed maximum duration for Durvalumab treatment. Treatment with Durvalumab continues until the physician determines its benefit for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Describe real world data on PFS of patients treated with Durvalumab in stage III NSCLC in the EAP in Brazil | June of 2018

OTHER OUTCOMES:
- To describe Overall response rate, defined as the proportion of patients who have a partial or complete response to durvalumab therapy. | June of 2018
- To describe Overall survival at 3 years, defined as the time from start of durvalumab therapy to death from any cause. | June of 2018
- To describe the sequence of lines of treatment in patients which have disease progression after durvalumab. | June of 2018

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Núcleo de Oncologia da Bahia S.A, Salvador, Estado de Bahia
  - Instituto Mário Penna, Belo Horizonte, Minas Gerais
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Postmus PE, Kerr KM, Oudkerk M, Senan S, Waller DA, Vansteenkiste J, Escriu C, Peters S; ESMO Guidelines Committee. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv1-iv21. doi: 10.1093/annonc/mdx222. No abstract available. PMID 28881918
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] De Ruysscher D, Botterweck A, Dirx M, Pijls-Johannesma M, Wanders R, Hochstenbag M, Dingemans AM, Bootsma G, Geraedts W, Simons J, Pitz C, Lambin P. Eligibility for concurrent chemotherapy and radiotherapy of locally advanced lung cancer patients: a prospective, population-based study. Ann Oncol. 2009 Jan;20(1):98-102. doi: 10.1093/annonc/mdn559. Epub 2008 Aug 20. PMID 18718891
- [Derived] Zukin M, Gondim V, Shimada AK, Lima EMEA, Mathias C, Barra WF, William Junior WN, Padoan M, Bittencourt Y, Yamamura R, Silva CEB, Rossato LJ, Monteiro CA, Jesus RG, Gossling G, Gelatti ACZ. Durvalumab as consolidation therapy in patients who received chemoradiotherapy for unresectable stage III NSCLC: Real-world data from an expanded access program in Brazil (LACOG 0120). J Bras Pneumol. 2025 Jan 13;50(6):e20240228. doi: 10.36416/1806-3756/e20240228. eCollection 2025. PMID 39813498